CLINICAL TRIAL: NCT00626509
Title: Sunitinib Either Before or After Cytoreductive Nephrectomy in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Sunitinib Before or After Surgery in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Carcinoma Renale (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GICR-GIR-1; CDR0000588423 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2007-005977-67
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: sunitinib malate
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any tumor cells that remain after surgery. It is not yet known whether sunitinib is more effective when given before or after surgery in treating kidney cancer.

PURPOSE: This randomized phase II trial is studying the side effects of sunitinib and to compare how well it works when given before or after surgery in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the activity of sunitinib malate when administered before vs after cytoreductive nephrectomy, in terms of response rate, in patients with metastatic renal cell carcinoma.
* To compare the safety of these regimens in these patients.

Secondary

* To compare the time to progression in patients treated with these regimens.
* To compare the duration of response in patients treated with these regimens.
* To compare the overall survival of patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo cytoreductive nephrectomy. Patients then receive adjuvant therapy comprising oral sunitinib malate once daily for 4 weeks. Treatment repeats every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Some patients may continue treatment beyond 1 year at the discretion of the investigator.
* Arm II: Patients receive neoadjuvant therapy comprising oral sunitinib malate once daily for 4 weeks. Treatment repeats every 6 weeks for 2 courses. After completion of neoadjuvant therapy, patients undergo cytoreductive nephrectomy followed by adjuvant sunitinib malate as in arm I.

After completion of study therapy, patients are followed every 2 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Proven metastatic renal cell carcinoma
* Measurable disease (according to RECIST criteria)
* Eligible for cytoreductive nephrectomy

  * Primary tumor is considered amenable to surgical extirpation by the attending surgeon
  * Thrombosis of the inferior vena cava below the epathic veins allowed
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Adequate hematology and coagulation
* Amylase and lipase normal
* Adequate hepatic, renal, and cardiac function
* Not pregnant
* Negative pregnancy test
* No uncontrolled hypertension and/or clinically significant cardiovascular events or disease within the past 12 months
* No other cancer within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* No prior early nephrectomy due to clinical condition
* No prior systemic therapy for renal cell carcinoma (e.g., chemotherapy, hormonal therapy, interferon, interleukin-2, lymphocyte-activated killer cells, or other biological response modifiers)
* More than 12 days since prior potent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * St. John's wort
  * Efavirenz
  * Tipranavir
* More than 7 days since prior potent CYP3A4 inhibitors, including any of the following:

  * Ketoconazole
  * Itraconazole
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * Delavirdine
  * Indinavir
  * Saquinavir
  * Ritonavir
  * Atazanavir
  * Nelfinavir
* No other concurrent approved or investigational anticancer treatment, including chemotherapy, biological response modifiers, hormonal therapy, or immunotherapy
* No concurrent participation in any other treatment clinical trial
* No concurrent palliative radiotherapy or surgery
* No concurrent drugs with proarrhythmic potential, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* Concurrent bisphosphonate therapy for metastatic bone disease allowed provided therapy was initiated at least 4 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Overall objective tumor response rate (complete response, partial response, stable disease, and progressive disease) as assessed by RECIST criteria
Adverse events as assessed by NCI CTCAE v3.0

SECONDARY OUTCOMES:
Time to progression
Duration of response
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Marco Venturini, MD, Principal Investigator — Ospedale Sacro Cuore
Locations (1):
- Ospedale Sacro Cuore, Negrar, Italy